CLINICAL TRIAL: NCT01638845
Title: Hip Fracture and Perineural Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008/072/HP
Record Dates: First submitted 2012-06-22; First posted 2012-07-12 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous perineural catheter (Active Comparator)
  Interventions: Procedure: continuous perineural catheter
- Control (No Intervention)

INTERVENTIONS:
Procedure: continuous perineural catheter — continuous perineural catheter
  Arms: continuous perineural catheter

SUMMARY:
INTRODUCTION: Hip Fracture is a public health problem because of its constantly increasing frequency and its high morbidity and mortality. The leading cause of death is cardiovascular decompensation, caused by painful phenomena associated with fracture and orthopedic surgery.With hip fracture, epidural local analgesia techniques have proven their benefit in mortality but are associated with numerous side effects that prevent routine use. Peripheral analgesic techniques locoregional the lumbar plexus, much safer, cause a decrease in postoperative pain after surgery for hip fracture and a decrease in mortality at 6 months. Elderly patients suffering from a hip fracture, no study has investigated the effect of local analgesia continuous femoral perineural catheter on the incidence of cardiovascular events in the perioperative period.

OBJECTIVE: The main objective of this work is to show that perineural analgesia block continuous local anesthetic reduces the incidence of cardiovascular complications in the preoperative period of a patient with a hip fracture and fact, show that this technique decreases the incidence of mortality at one year of patients with a hip fracture (secondary objective).

MATERIAL AND METHODS: This is a prospective, multicenter, randomized, descriptive type. It compares two populations of patients: one has a perineural analgesia by continuous infusion via a catheter of ropivacaine (n = 157) associated with a systemic analgesia and the other only systemic analgesia without development of a catheter perineural (n = 157). The duration of patient participation will be 12 months. In the first 24 hours after a hip fracture after randomization, study participants will benefit from the installation under strict asepsis, a continuous block by catheter, placed by an anesthesiologist experienced control room post-interventional. The local analgesia will be provided by continuous administration via the perineural catheter, ropivacaine for 5 days for the treated group. Except the local analgesia protocol, the protocols pre-and postoperative systemic analgesia and general anesthesia will be identical for all participants of the 2 groups, similar to techniques proposed in the context of everyday clinical practice, ensuring analgesia optimal for all patients in the study. The main features will be found three bioassays Troponin IC and 3 electrocardiograms at the entrance to the hospital, J3 and J5 after inclusion. In addition, cardiovascular clinical monitoring and quantification of pain ( will be performed daily for 8 days after inclusion. Finally, an assessment of higher functions by ladder MMS will be conducted at the entrance, J3, J5 and J8. Moreover, a survey of survival at 1 month, 3 months and 1 year will be realized.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an age greater than or equal to 60 years
* Patients who have written, informed consent was obtained
* Patients evaluated ASA 1, 2 and 3 according to the classification of the American Society of Anesthesiologists (detailed below)
* Patients undergoing surgery for hip fracture
* Time less than 24 hours after a hip fracture

Exclusion Criteria:

* cons indication to regional anesthesia (constitutional or acquired disorder of coagulation, sepsis, local infection of the puncture area, history of vascular surgery prosthetic femoral neuropathy scalable, allergy to local anesthetics)
* weight <40Kg
* Patients receiving treatment hypocoagulable or antiplatelet therapy of type dipyridamole, ticlopidine and platelet αIIbβ3 receptor antagonists (excluding aspirin and clopidogrel)
* cons-indication for standardized anesthetic technique in this study
* cons-indication for analgesics used postoperatively (respiratory failure, severe liver failure, brain injury associated with intracranial hypertension, uncontrolled epilepsy, simultaneous treatment with MAOIs, hypersensitivity to opioids)
* Patient unable to give informed consent
* adults under guardianship or curator
* persons not affiliated with a health insurance plan
* A person deprived of liberty

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with cardiovascular events during the preoperative period | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Vincent COMPERE, Pr, Principal Investigator — UH Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043